CLINICAL TRIAL: NCT06626568
Title: Comparison Between Ultrasound Guided Subacromial and Systemic Injection of Steroid for Frozen Shoulder: a Double Blind Multicenter Pilot Study for Randomized Control Trial
Brief Title: Comparison of Ultrasound-Guided Subacromial vs. Systemic Steroid Injections for Frozen Shoulder: a Multicenter Pilot Study
Acronym: CUSIS-FS-Pilot
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-0405
Record Dates: First submitted 2024-09-29; First posted 2024-10-04 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2024-09

CONDITIONS: Frozen Shoulder
Keywords: frozen shoulder; intramuscular injection; subacromial injection; compound betamethasone; ultrasound guidance
MeSH Terms: conditions — Bursitis | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- gluteal injection (Experimental): gluteal injection of 1 ml of Compound betamethasone and 4 ml of normal saline at week 0,2,4, ultrasound-guided subacromial injection of 5 ml of normal saline at week 0,2,4.
  The participants were instructed to perform home rehabilitation exercise for 12 weeks. 30 minutes of home-based self-rehabilitation exercises in the morning, afternoon, and evening, with a total of 90 minutes per day. Standard instructional videos and demonstrations by outpatient rehabilitation therapists are provided to participants. Each exercise, including wall-climbing, table-climbing, and back-climbing, should be performed for 10 minutes, with a total of 30 minutes per session.
  Interventions: Drug: Compound betamethasone Injection(Gluteal muscle injection); Other: Normal Saline as Placebo (ultrasound-guided subacromial injection); Behavioral: home exercise
- subacromial injection (Active Comparator): gluteal injection of 5 ml normal saline at week 0,2,4, ultrasound-guided subacromial injection of 1 ml of Compound betamethasone and 4 ml of normal saline at week 0,2,4.
  The participants were instructed to perform home rehabilitation exercise for 12 weeks. 30 minutes of home-based self-rehabilitation exercises in the morning, afternoon, and evening, with a total of 90 minutes per day. Standard instructional videos and demonstrations by outpatient rehabilitation therapists are provided to participants. Each exercise, including wall-climbing, table-climbing, and back-climbing, should be performed for 10 minutes, with a total of 30 minutes per session.
  Interventions: Drug: Compound betamethasone Injection(Subacromial Ultrasound Guided injection); Other: Normal Saline as Placebo (gluteal muscle inection); Behavioral: home exercise

INTERVENTIONS:
Drug: Compound betamethasone Injection(Gluteal muscle injection) — gluteal injection of 1 ml of Compound betamethasone and 4 ml of normal saline at week 0,2,4
  Arms: gluteal injection
Drug: Compound betamethasone Injection(Subacromial Ultrasound Guided injection) — ultrasound-guided subacromial injection of 1 ml of Compound betamethasone and 4 ml of normal saline at week 0,2,4.
  Arms: subacromial injection
Other: Normal Saline as Placebo (ultrasound-guided subacromial injection) — ultrasound-guided subacromial injection of 5 ml of normal saline at week 0,2,4.
  Arms: gluteal injection
Other: Normal Saline as Placebo (gluteal muscle inection) — gluteal injection of 5 ml normal saline at week 0,2,4.
  Arms: subacromial injection
Behavioral: home exercise — The participants were instructed to perform home rehabilitation exercise for 12 weeks. 30 minutes of home-based self-rehabilitation exercises in the morning, afternoon, and evening, with a total of 90 minutes per day. Standard instructional videos and demonstrations by outpatient rehabilitation therapists are provided to participants. Each exercise, including wall-climbing, table-climbing, and back-climbing, should be performed for 10 minutes, with a total of 30 minutes per session.

SUMMARY:
The goal of this multicenter pilot study is to validate the effectiveness of extending the injection interval between betamethasone doses from one to two weeks for treating frozen shoulder (adhesive capsulitis) in adults aged 18 to 75. This study also aims to screen potential study centers and gather data to refine the sample size calculation for a larger, future trial. The main questions it aims to answer are:

* Does extending the interval between injections maintain effectiveness in improving shoulder function and reducing pain for frozen shoulder?
* Which centers in this pilot study are qualified for a larger, future trial?
* What is the appropriate sample size for conducting a multicenter RCT study with the same research design at the selected centers?

Participants will:

* Receive 3 injections over 4 weeks and will be followed up for another 8 weeks
* Complete shoulder function assessments
* Perform home rehabilitation exercises

ELIGIBILITY:
Inclusion Criteria:

1. History of ≤9 months, clinically diagnosed with primary frozen shoulder (including frozen shoulder associated with diabetes).
2. Aged between 18 and 75 years old
3. Pain NRS score ≥4
4. Measured passive range of motion of the affected shoulder in at least two of the three directions (forward flexion, external rotation with arm at the side, and internal rotation with arm at the side) is reduced by 25% or more compared to the contralateral normal shoulder.
5. Exclusion of osteoarthritis, dislocation, and other shoulder abnormalities through X-ray and MRI of the affected shoulder.

Exclusion Criteria:

1. Secondary frozen shoulder caused by thyroid disease, cardiovascular disease, cancer, stroke, radiotherapy, neurosurgery, or breast surgery (excluding diabetes); secondary frozen shoulder caused by major shoulder trauma requiring medical care (e.g., fractures, dislocations, rotator cuff tears).
2. Full-thickness rotator cuff tear in the affected shoulder confirmed by MRI (excluding rotator cuff tendinopathy and partial-thickness rotator cuff tear in patients with frozen shoulder without a history of major shoulder trauma).
3. Patients unable to undergo MRI due to financial reasons, claustrophobia, pacemaker, or other metallic implants in the body.
4. Local infection in the affected shoulder or other contraindications to shoulder injections.
5. Patients with contraindications to steroid therapy (e.g., poorly controlled blood sugar in diabetes).
6. Patients with frozen shoulder who have already undergone shoulder injections, manipulation under anesthesia, arthroscopic capsular release, or open surgery for capsular release.
7. Received any form of steroid treatment within the past 3 months.
8. History of glucocorticoid use for more than 3 months.
9. Bilateral frozen shoulder or a history of frozen shoulder in the contralateral shoulder.
10. Pregnant or breastfeeding women.
11. Patients lacking the cognitive ability to comply with the study protocol.
12. Patients not residing in the area where the study is being conducted.
13. Patients with compensation claims or legal disputes related to workplace injury or car accidents.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-08-21 (Actual); Study Completion 2025-09-02 (Actual)

PRIMARY OUTCOMES:
Shoulder Pain and Disability Index (SPADI) | Baseline and 12 weeks
  The SPADI score ranges from 0 to 100. A score of 0 indicates no pain or disability, while a score of 100 reflects the worst possible pain and maximum functional disability in the shoulder.
  Data entry will be performed by blinded research staff. They will present the paper CRF sample form to the participants and ask questions one by one, directly entering the responses of participants into the corresponding electronic CRF form in the EDC system using handheld electronic devices (such as smartphones, tablets, or laptops).

SECONDARY OUTCOMES:
progression rate of rotator cuff tears | From enrollment to the end of follow-up at 12 weeks
  Third-party experts will conduct blinded readings of shoulder MRI scans, classifying rotator cuff status into three grades: Grade I (intact), Grade II (partial tear), and Grade III (complete tear). Patients classified as Grade III at week 0 will be excluded from the study, as baseline grading (determined by each research center) assesses eligibility per exclusion criterion 2. The lead center provided MRI reading training to all centers, using T2-weighted images with a pure white fluid signal occupying full or partial thickness of the rotator cuff across at least two consecutive MRI slices as the diagnostic criterion for full- or partial-thickness tears. Patients with Grade I or II tears at week 0 will receive study treatment and be followed up at week 12. Tear progression is defined as an increase of at least one grade between weeks 0 and 12, assessed by blinded experts. The progression rate is the number of subjects with progression divided by the total number in each group.
short version of Disabilities of the Arm, Shoulder, and Hand Questionnaire (QuickDASH） | Baseline and 12 weeks
  The QuickDASH score ranges from 0 to 100. A score of 0 means no disability, and a score of 100 signifies the highest level of disability related to arm, shoulder, and hand function.
  Data entry will be performed by blinded research staff. They will present the paper CRF sample form to the participants and ask questions one by one, directly entering the responses of participants into the corresponding electronic CRF form in the EDC system using handheld electronic devices (such as smartphones, tablets, or laptops).
Numerical Rating Scale (NRS) | Baseline and 12 weeks
  The NRS score ranges from 0 to 10. A score of 0 indicates no pain, while a score of 10 reflects the worst possible pain.
  Data entry will be performed by blinded research staff. They will present the paper CRF sample form to the participants and ask questions one by one, directly entering the responses of participants into the corresponding electronic CRF form in the EDC system using handheld electronic devices (such as smartphones, tablets, or laptops).
five-level EuroQol five-dimensional questionnaire (EQ-5D-5L) | Baseline and 12 weeks
  The EQ-5D-5L provides an overall health utility score ranging from -0.281 to 1, where 1 represents perfect health, zero represents a state equivalent to death, and negative values indicate health states worse than death.
  It also reports on five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each rated on five levels from no problems to extreme problems.
  Data entry will be performed by blinded research staff. They will present the paper CRF sample form to the participants and ask questions one by one, directly entering the responses of participants into the corresponding electronic CRF form in the EDC system using handheld electronic devices (such as smartphones, tablets, or laptops).
passive range of motion of shoulder | Baseline and 12 weeks
  The passive range of motion for shoulder flexion, abduction, internal rotation (at the side), and external rotation (at the side) on the affected side will be measured using a goniometer by trained researchers following a pre-established standard operating procedure.
Direct Medical Cost | Baseline
  The costs of healthcare resources used for the diagnosis and treatment of frozen shoulder of the participant, including medication fees, medical expenses, testing fees, nursing fees and hospitalization costs. The questionnaire surveys the cost by the participant since the onset of frozen shoulder.
Direct Medical Cost | Baseline and week2
  The costs of healthcare resources used for the diagnosis and treatment of frozen shoulder of the participant, including medication fees, medical expenses, testing fees, nursing fees and hospitalization costs. The questionnaire surveys the cost by the participant since the last outpatient research follow-up.
Direct Medical Cost | Week2 and week4
  The costs of healthcare resources used for the diagnosis and treatment of frozen shoulder of the participant, including medication fees, medical expenses, testing fees, nursing fees and hospitalization costs. The questionnaire surveys the cost by the participant since the last outpatient research follow-up.
Direct Medical Cost | Week4 and week8
  The costs of healthcare resources used for the diagnosis and treatment of frozen shoulder of the participant, including medication fees, medical expenses, testing fees, nursing fees and hospitalization costs. The questionnaire surveys the cost by the participant since the last outpatient research follow-up.
Direct Medical Cost | Week8 and week12
  The costs of healthcare resources used for the diagnosis and treatment of frozen shoulder of the participant, including medication fees, medical expenses, testing fees, nursing fees and hospitalization costs. The questionnaire surveys the cost by the participant since the last outpatient research follow-up.
work absenteeism | Week 0
  The questionnaire surveys the number of workdays missed since the onset of frozen shoulder is collected at baseline.
work absenteeism | Week 0 and Week 2
  The questionnaire surveys the number of workdays missed by the subject since the last outpatient research follow-up.
work absenteeism | Week 2 and Week 4
  The questionnaire surveys the number of workdays missed by the subject since the last outpatient research follow-up.
work absenteeism | Week 4 and Week 8
  The questionnaire surveys the number of workdays missed by the subject since the last outpatient research follow-up.
work absenteeism | Week 8 and Week 12
  The questionnaire surveys the number of workdays missed by the subject since the last outpatient research follow-up.
Unplanned concomitant use of analgesics | Week 2
  This questionnaire surveys the usage of unplanned concomitant analgesic medications by the subject since the last outpatient research follow-up.
Unplanned concomitant use of analgesics | Week 4
  This questionnaire surveys the usage of unplanned concomitant analgesic medications by the subject since the last outpatient research follow-up.
Unplanned concomitant use of analgesics | Week 8
  This questionnaire surveys the usage of unplanned concomitant analgesic medications by the subject since the last outpatient research follow-up.
Unplanned concomitant use of analgesics | Week 12
  This questionnaire surveys the usage of unplanned concomitant analgesic medications by the subject since the last outpatient research follow-up.
Glycated Hemoglobin (HbA1c) | week 0 and week 12
  Depending on the specific assay methods used by the laboratory departments of different study centers, HbA1c will be measured by high-Performance Liquid Chromatography (HPLC), Immunoturbidimetric Method, Enzymatic Method, Affinity Chromatography, Electrophoresis, Capillary Electrophoresis or Ion-Exchange Chromatography.
glycated albumin | week 0 and week 4
  Depending on the specific assay methods used by the laboratory departments of different study centers, glycated albumin will be measured by Enzymatic Method, Immunoturbidimetric Method, High-Performance Liquid Chromatography (HPLC), Affinity Chromatography, or Immunoelectrophoresis.

OTHER OUTCOMES:
incidence of serious adverse events (SAE) | From enrollment to the end of follow-up at 12 weeks
  The incidence of serious adverse events (SAE) at 12 weeks
incidence of adverse events (AE) | From enrollment to the end of follow-up at 12 weeks
  The incidence of adverse events (AE) at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bin Han, Medical Doctor, Principal Investigator — The 2nd Affiliated Hospital of Zhejiang University
Locations (9):
- China (9):
  - Guangde County People's Hospital, Xuancheng, Anhui
  - Yangpu District Central Hospital of Shanghai, Shanghai, Shanghai Municipality
  - Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - The First People's Hospital of Linping District, Hangzhou, Hangzhou, Zhejiang
  - Huzhou Central Hospital, Huzhou, Zhejiang
  - Pujiang People's Hospital, Jinhua, Zhejiang
  - First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang
  - Xiangshan County Traditional Chinese Medicine Hospital Healthcare Group, Ningbo, Zhejiang
  - Shengzhou People's Hospital, Shanhu, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
The current registration is for a pilot study for a later larger trial. We will consider sharing the data after the completion of the subsequent full trial.
Supporting Information: Study Protocol, ICF
Time Frame: We will consider sharing the data after the completion of the subsequent full trial.
Access Criteria: Researchers who have published at least one peer-reviewed clinical study on frozen shoulder, as well as journal editors and corresponding peer reviewers involved in reviewing our subsequent formal study (CUSIS-FS, a multicenter RCT on frozen shoulder), will be able to access the IPD and supporting information.